CLINICAL TRIAL: NCT00811031
Title: A Phase II Study of Pre-operative Docetaxel for Progressive Localized Castration Resistant Prostate Cancer
Brief Title: Preoperative Docetaxel for Localized Progressive Castration-resistant Prostate Cancer (CRPC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0045
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Prostate Cancer
Keywords: Prostate; prostate gland; prostate cancer markers; Taxotere®; Docetaxel; Prednisone; Castration Resistant Prostate Cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Taxotere + Prednisone (Experimental)
  Interventions: Drug: Taxotere; Drug: Prednisone

INTERVENTIONS:
Drug: Taxotere — 75 mg/m^2 Day 1 of every 21-day cycle by vein for 4 cycles prior to surgery.
  Other Names: docetaxel
Drug: Prednisone — 5 mg twice a day by mouth.

SUMMARY:
Objectives:

Primary:

* To evaluate the association of the probability of increase in phosphorylation of platelet-derived growth factor receptor (PDGFR) of > 0.5 in peripheral blood leucocytes following pre-operative docetaxel chemotherapy, with progression-free survival in localized castration-resistant prostate cancer (CRPC)

Secondary:

* To evaluate the association of the probability of increase in phosphorylated platelet-derived growth factor receptor (PDGFR) expression in peripheral blood leucocytes > 0.5 with indices of tumor regression including PSA-decline by 50% and measures of objective regression of tumor by transrectal MRI following pre-operative docetaxel therapy.
* Explore associations of probability of increase in phosphorylated PDGFR in peripheral blood leucocytes following pre-operative docetaxel therapy with plasma PDGF kinetics and spatial and quantitative PDGF and phosphorylated PDGFR expression in tumor and stromal compartments in resected specimens.
* Evaluate the association of probability of increase in phosphorylated PDGFR expression in peripheral blood leucocytes following pre-operative docetaxel chemotherapy with overall survival outcomes.
* Assess global quality of life measures at baseline and 6 and 12 months post-operatively.
* Create a tissue archive comprising tumor and peripheral blood specimens as a suitable resource for future genomic and proteomic studies.

DETAILED DESCRIPTION:
The Study Drugs:

Docetaxel is designed to stop the growth of cancer cells, which may cause the cells to die. It is believed to be weakly effective at killing blood vessels in cancer cells as well.

Prednisone and docetaxel are commonly used to treat prostate cancer.

Study Drug Administration:

If you are found to be eligible to take part in this study, on Day 1 of every 21-day study "cycle", you will receive docetaxel through a needle in your vein over 1 hour.

Everyday, you will take prednisone by mouth 2 times a day (in the morning and evening). You should take prednisone with meals.

You will take dexamethasone by mouth at 12 hours and 6 hours before you receive docetaxel. This is to help reduce the risk of any allergic reaction and fluid retention. It is important that you take this drug on schedule.

Study Visits:

On Day 1 of each cycle, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight.
* Your performance status will be recorded.
* You will be asked about any drugs or treatments you may be receiving.
* You will be asked about any side effects you have experienced since your last visit.

Blood (about 2 teaspoons) will be drawn for routine tests and to test for PSA and testosterone levels.

On Day 1 of Cycle 3, blood (about 2 teaspoons) will be drawn to test for PDGFR and PDGF levels.

Surgery:

If you complete 2 cycles or more, you will be eligible to have surgery as part of this study.

If you are eligible, no more than 21 days after your last dose of docetaxel, you will have surgery to remove your prostate gland. You will sign a separate consent for this surgery, which will describe the procedure and its risks in detail.

Before surgery, probably at your pre-surgical visit, blood (about 2 teaspoons) will be drawn to test for PDGFR and PDGF levels.

Length of Study:

You will take the study drug for up to 4 cycles before having surgery. You will be off study treatment after you have surgery. You will be taken off study early if you experience intolerable side effects or the disease gets worse.

This is an investigational study. Docetaxel given with prednisone is commercially available and FDA approved for the treatment of prostate cancer.

Up to 28 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with adenocarcinoma of the prostate (ductal or acinar).
2. Symptomatic or evidence of progressive disease in the primary tumor by digital rectal examination, cystoscopy and/or radiological imaging without symptomatic or objective evidence of systemic disease progression.
3. Patients must have a castrate serum testosterone level (</= 50ng/ml) documented in the last six weeks. For patients who are medically castrated, luteinizing hormone releasing hormone analog must continue to maintain testicular suppression.
4. Patients on antiandrogens should be discontinued from flutamide, nilutamide or cyproterone acetate for at least 4 weeks and bicalutamide for 6 weeks. If localized progression is documented during or after this time interval, patients are eligible. Patients who have not had response to deferred (secondary) therapy with antiandrogens do not have to satisfy this waiting period prior to enrollment.
5. Surgically resectable disease as assessed by the collaborating urological oncologist.
6. Patients must be >/= 18 years of age.
7. Patients must have a performance status of </= 2 (ECOG).
8. Patients must have an expected survival from cancer or co-morbidity of six months.
9. Patients will not receive any concurrent biological, immunological, second-line hormonal therapy or chemotherapy. Patients receiving replacement or therapeutic doses of corticosteroid for non-malignant disease while disease progression was established may continue on such therapy.
10. Patients may not have received docetaxel or other chemotherapeutic agents in the last 6 months or have been defined as docetaxel-resistant or intolerant previously.
11. Patients must have adequate bone marrow function defined as an Hgb >/= 8.0 g/dl, absolute peripheral granulocyte count of >/= 1,500/mm^3 and platelet count of >/= 100,000/mm^3.
12. Patients must have adequate hepatic function defined with a bilirubin of </= upper limits of normal. AST and ALT and Alkaline Phosphatase must be within the range allowing for eligibility. In determining eligibility the more abnormal of the two values (AST or ALT) should be used (see chart below in Study Plan).
13. Patients must have adequate renal function defined as creatinine clearance >/= 30 cc/min (measured or calculated by Cockcroft and Gault formula).
14. Must be fully recovered from any previous surgery, in terms of wound healing.
15. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of the institution.
16. Men with the ability to father a child must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

Exclusion Criteria:

1. Patients with severe or uncontrolled infection defined as symptomatic and/or requiring intravenous antibiotics.
2. Patients with small cell or sarcomatoid variant of prostate cancer.
3. Patients with symptomatic congestive heart failure (CHF), pulmonary embolus, vascular thrombosis, transient ischemic attack, cerebrovascular accident, unstable angina or MI in the last 6 months or evidence of active myocardial ischemia by symptoms or ECG.
4. Oxygen-dependent lung disease, > grade 2 peripheral neuropathy, uncontrolled hypertension or uncontrolled diabetes mellitus.
5. Active second malignancies. Non-threatening second malignancies such as superficial low-grade transitional cell carcinoma of the bladder, Rai Stage 0 chronic lymphocytic leukemia or stable small renal cell carcinomas may be exempt from such stipulation at the discretion of the Principal Investigator.
6. Patients who are unwilling to provide blood or tissue specimens required for the primary objectives of the study.
7. Overt psychosis or mental disability or otherwise incompetent to give informed consent. Patients with a history of non-compliance with medical regimens or who are considered potentially unreliable.
8. Patients with a history of severe hypersensitivity reaction to Taxotere® or other drugs formulated with polysorbate 80.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Pre-to-post chemotherapy increase phosphorylation of platelet-derived growth factor receptor (PDGFR) | PDGFR will be estimated for each patient based on blood samples taken at day 0 and at day 42 using the Bayesian survival time regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Lance Pagliaro, MD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org